CLINICAL TRIAL: NCT03358927
Title: Immediate Fast-Track Versus Standard Care for Persons Living With HIV in Haiti: A Randomized Pilot Study
Brief Title: Immediate Fast-Track Versus Standard Care for Persons Living With HIV in Haiti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other); Weill Medical College of Cornell University (Other); Duke University (Other); Florida International University (Other); Analysis Group, Inc. (Industry)
Responsible Party: Principal Investigator, Serena Patricia Koenig, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH114739 (NIH)
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Fast-track care; Behavioral economics; Differentiated care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Group (Active Comparator): Deferred fast-track care
  Interventions: Behavioral: Deferred Fast-Track Care
- Immediate Fast-Track Group (Experimental): Immediate fast-track care
  Interventions: Behavioral: Immediate Fast-Track Care

INTERVENTIONS:
Behavioral: Immediate Fast-Track Care — Eligible for fast-track care at enrollment
  Arms: Immediate Fast-Track Group
Behavioral: Deferred Fast-Track Care — Eligible for fast-track care after 6 months on ART
  Arms: Standard Group

SUMMARY:
In the proposed R34 grant, the investigators will develop and test a strategy of immediate fast-track care. The study population will include adult patients with early HIV infection. Participants will be randomized to immediate fast-track or standard (deferred fast-track) care. All participants will receive same-day HIV testing and ART initiation prior to study enrollment. The intervention group will receive immediate fast-track care, which is conditional upon timely visits, and after 24 weeks in care, an undetectable viral load (HIV-1 RNA <200 copies/ml). The standard group will be eligible to start fast-track care at 24 weeks, if they are on time for that visit and have an undetectable viral load. Participants in either group who are >3 days late for any fast-track visit will lose fast-track care for that visit; those in either group with detectable viremia on their 24-week viral load test will be evaluated by a physician, with follow-up visits every 4 weeks until they have an undetectable viral load. Participants will be followed for 48 weeks. With the proposed pilot study, the investigators aim to conduct the formative work that is necessary to successfully implement a future clinical trial with the same primary outcome. The investigators hypothesize that immediate fast-track care will result in higher retention with viral suppression.

DETAILED DESCRIPTION:
This study is a randomized, open-label pilot study comparing immediate fast-track vs. standard care for patients with WHO Stage 1 or 2 disease at HIV diagnosis. Participants will be enrolled on the day of HIV diagnosis, and will be followed for 48 weeks. The total sample size will be 254 participants; of these, 56 will be patients or providers enrolled in one-time focus groups, 20 will be enrolled for testing the manuals and study procedures, and 178 will be enrolled in the pilot RCT.

The study site is GHESKIO (Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic Infections) in Port-au-Prince, Haiti. The study population includes men and women who are at least 18 years of age who are ART-naïve, and who present with WHO Stage 1 or 2 diseases at HIV diagnosis.

Participants in both groups will initiate ART on the day of HIV testing, prior to enrollment and randomization. They will then be randomized to immediate versus standard (deferred fast-track) care. Those in the immediate group will start fast-track care on the day of HIV testing. Those in the standard group will start fast-track care if they are on time for their 24-week visit, with HIV-1 RNA <200 copies/ml. Participants in both groups will receive identical care from weeks 24 to 48.

Once a patient qualifies for fast-track care, it is provided in the same manner for both groups.

* Reminder phone call and point-of-service dispensing of ART: The CHW calls patient one day in advance, to ensure they can attend visit. If patient responds in the affirmative, then their ART and prophylactic medications are packaged in advance.
* Minimal waiting time to see clinician, with short, focused visits: Total visit time is about 30 minutes.
* Less frequent clinic visits: Other than the first 3 months for the immediate group, fast-track care includes quarterly nurse visits, with CHW phone calls during months when no clinic visit is scheduled;
* Nurse-led care: Fast-track visits are all staffed by nurses, except in the case that a patient has a new symptom; in that case, the patient receives a fast-track physician evaluation, with appropriate fast-track follow-up care. For example, in the rare case that a patient develops active TB, they will receive fast-track care with physician and nurse visits as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of ≥18 years of age
* Ability and willingness to give written informed consent
* Documentation of positive HIV status (test conducted at GHESKIO), and initiation of same-day ART prior to enrollment
* Physician-confirmed WHO Stage 1 or 2 disease
* Acceptance of HIV diagnosis, defined as affirmative responses to two questions: "I believe that HIV and AIDS exist" and "I believe that the results of my HIV test show that I am infected".
* Access to a phone, or able to provide a contact person with a phone (this does not require disclosure of HIV status to the contact person)
* Agreement to provide a contact phone number and address, and to accept home visits from a CHW.

Exclusion Criteria:

* Any use of ART in the past
* Pregnancy or breastfeeding at the screening visit
* WHO Stage 3 or 4 disease
* Active drug, alcohol use, or mental condition that would interfere with the ability to adhere to study requirements, in the opinion of the study physician
* Score of <3 for any of the 7 questions on the ART readiness survey
* Planning to transfer care to another clinic during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Viral Suppression; cut-off <200 copies/ml | 48 weeks after enrollment
  HIV-1 RNA <200 copies/ml

SECONDARY OUTCOMES:
Viral Suppression; cut-off <50 copies/ml | 48 weeks after enrollment
  HIV-1 RNA <50 copies/ml
Viral Suppression; cut-off <1000 copies/ml | 48 weeks after enrollment
  HIV-1 RNA <1000 copies/ml
Adherence by pharmacy refill records | 48 weeks after enrollment
  ART dispensed by the pharmacy for at least 90% of the days in the study period (302 days of ART dispensed during the 336-day study period)
Cost-effectiveness | 48 weeks after enrollment
  Cost per patients with undetectable viral load
Connectedness to Treatment Setting Scale | Day of enrollment, and 24 weeks and 48 weeks after enrollment
  Mean score; range 10-60; a higher score indicates greater connection to treatment setting
State Hope Scale | Day of enrollment, and 24 weeks and 48 weeks after enrollment
  Mean score; range 6 to 30; a higher score indicates greater hopefulness
Patient Satisfaction Survey | Weeks 2, 24, and 48 after enrollment
  Mean score; range 5 to 25; a higher score indicates greater satisfaction
Social Provisions Scale | Day of enrollment, and 24 and 48 weeks after enrollment
  Mean score; range 24 to 96; a higher score indicates greater degree of perceived support
Coping Survey | Weeks 2, 24, and 48 after enrollment
  Mean score; range 38 to 152; a higher score indicates a greater sense of being able to cope with a situation

CONTACTS AND LOCATIONS:
Overall Officials: Serena Koenig, MD, Principal Investigator — Brigham and Women's Hospital/GHESKIO; Jean Pape, MD, Study Director — GHESKIO; Weill Medical College of Cornell University
Locations (1):
- GHESKIO, Port-au-Prince, Haiti

IPD SHARING:
Plan to Share IPD: Yes
We will post an anonymized dataset after the study is complete.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available at the time of publication of the primary study results.
Access Criteria: Information will be posted online.